CLINICAL TRIAL: NCT02389543
Title: A Multi-Center, Phase 1/2, Open-Label Study of Selinexor (KPT- 330), Lenalidomide, and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Selinexor (KPT- 330), Lenalidomide, & Dexamethasone in Relapsed/Refractory Multiple Myeloma Patients
Acronym: SLAM
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated this trial and added a Lenalidomide arm to KCP-330-017
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-011
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: KPT-330; Selinexor; Multiple Myeloma; Relapsed/refractory; Lenalidomide; Dexamethasone; Karyopharm
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — selinexor; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Selinexor (1x/week), Lenalidomide, & Dexamethasone (Experimental): Lenalidomide will be dosed initially at 15 mg daily, and if that dose is tolerated per dose-limiting toxicity (DLT criteria,) it will be increased to 25 mg for that arm. Selinexor will be started at 80 mg (~45 mg/m2) once weekly in combination with dexamethasone 40 mg once weekly with each dose of selinexor. If the selinexor 80 mg dose is tolerated per DLT criteria, the dose will be increased to 100 mg (~60 mg/m2) and evaluated for MTD, tolerability and efficacy.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Dexamethasone
- B: Selinexor (2x/week), Lenalidomide, & Dexamethasone (Experimental): Lenalidomide will be dosed initially at 15 mg daily, and if that dose is tolerated per DLT criteria, it will be increased to 25 mg for that arm. Selinexor will be started at 60 mg (~35 mg/m2) twice weekly in combination with dexamethasone 20 mg twice weekly with each dose of selinexor; dexamethasone 20 mg will also be given, without selinexor, on Days 22 and 24. If the selinexor 60 mg dose is tolerated per DLT criteria, the dose will be increased to 80 mg (~45 mg/m2) and evaluated for MTD, tolerability and efficacy.
  Interventions: Drug: Selinexor; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Two different dosing schedules will be tested, once weekly and twice weekly. If the selinexor 80 mg dose is tolerated, the dose will be increased to 100 mg.
  Other Names: KPT-330
Drug: Lenalidomide — In both arms, lenalidomide will be started at 15 mg/day (Dose Level 1) and, if tolerated per DLT criteria, will be escalated to 25 mg/day (Dose Level 2).
Drug: Dexamethasone — Dexamethasone will be given in combination with each dose of selinexor on the once weekly treatment arm.
  For the twice weekly arm dexamethasone will be given in combination with each dose of selinexor and will also be given without selinexor on Days 22 and 24.

SUMMARY:
This is an open-label, randomized clinical study with two stages to assess the maximum tolerated dose (MTD), efficacy, and safety of selinexor, lenalidomide, and dexamethasone (SLd) in patients with relapsed/refractory (RR) multiple myeloma (MM). The stages are dose escalation (Phase 1) and expansion (Phase 2).

DETAILED DESCRIPTION:
In Phase 1 (Dose Escalation), patients will be randomized to either once-weekly (Arm A) or twice- weekly (Arm B) dosing with selinexor. Dose escalation will be performed within each arm for both lenalidomide and selinexor to determine the selinexor MTD for that arm. Each arm will be expanded until approximately 17 patients have been treated at the MTD in each arm. The Sponsor and Investigator will review the MTD, efficacy, and safety data from Phase 1 to determine which dose schedule (Arm A or B) to be used as the RP2D dose in the Expansion Phase.

In Phase 2 (Expansion), patients who had received the MTD dose that was nominated for RP2D will continue at the same dose. Patients who did not receive the RP2D for that arm will stay on their Phase 1 dose. Additional patients will be accrued, as needed, to achieve the target population size of approximately 34 patients at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis, measurable disease and evidence of disease progression of MM.
* Relapsed or refractory to the most recently received therapy. Relapsed is defined as documented evidence of PD after achieving at least SD for ≥ 1 cycle. Refractory disease is defined as ≤ 25% response (i.e., patients never achieved minimal response or better) or progression during therapy or within 60 days after completion of therapy.
* Symptomatic MM, based on IMWG guidelines. Patients must have measurable disease.

Exclusion Criteria:

* Smoldering MM.
* Multiple myeloma that does not express M-protein or FLC (i.e., non-secretory MM is excluded), and quantitative immunoglobulin levels cannot be used instead.
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome
* Active MM involving the central nervous system (CNS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) | 12 months
  Determine the maximum tolerated dose (MTD) of selinexor in the combination SLd in patients with RR MM, as determined by dose limiting toxicities (DLTs), efficacy, and safety
Overall response rate (ORR) | 12 months
  According to the International Myeloma Working Group [IMWG] criteria, Overall Response Rate (ORR) includes: stringent complete response [sCR], complete response [CR], very good partial response [VGPR], and partial response [PR]